CLINICAL TRIAL: NCT02738268
Title: Low-level Laser Therapy as a Tool for the Prevention of Radiodermatitis in Head and Neck Cancer Patients
Brief Title: Laser Therapy for the Prevention of Radiodermatitis in Head and Neck Patients
Acronym: DERMISHEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Prof. dr. Jeroen Mebis, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dermishead-001
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Head Cancer; Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Sham Comparator): Control group: receives sham laser (2x/week) in combination with standard skin care starting from day 1 of radiotherapy
  Interventions: Device: sham laser
- Treatment Group (Experimental): Treatment Group: receives low-level laser therapy (2x/week) in combination with standard skin care starting from day 1 of radiotherapy
  Interventions: Device: Low-level laser therapy

INTERVENTIONS:
Device: Low-level laser therapy — Low-Level Laser Therapy will be applied, twice a week, from the start of radiotherapy treatment in combination with the standard skin care.
  Other Names: LLLT
  Arms: Treatment Group
Device: sham laser
  Arms: Control group

SUMMARY:
Up to 90% of the radiotherapy patients will develop a certain degree of skin reaction at the treated area, also known as radiodermatitis (RD).

Currently, there is a wide variety of strategies to manage RD, including creams, gels, ointments, wound dressings. However, up to now, there is still no comprehensive, evidence-based consensus for the treatment of RD. Low-level laser therapy (LLLT) is a promising, non-invasive technique for treating RD. In a recent study conducted in our research group, LLLT prevented the aggravation of RD and provided symptomatic relief in patients undergoing radiotherapy for breast cancer after breast-sparing surgery. This was the first prospective study investigating the potential of LLLT for RD. In the current study, we want to investigate the efficacy of LLLT as a tool for the prevention of radiodermatitis in head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of head and neck squamous cell carcinomas (HNSCC) starting in the lip, salivary gland, oral cavity (mouth), nasal cavity (inside the nose), paranasal sinuses, pharynx, or larynx
* Scheduled for radiotherapy (>60 Gy), chemo-irradiation or bio-radiation either as primary or as post-operative treatment to the head and neck region
* Age ≥ 18 years
* Able to comply to the study protocol
* Able to sign written informed consent
* Signed written informed consent

Exclusion Criteria:

* Previous irradiation to the head and/or neck region
* Metastatic disease
* Patients with pre-existing skin rash, ulceration or open wound in the treatment area
* Patients with known allergic and other systemic skin diseases even when not directly affecting irradiated fields
* Substance abuse patients or patients with medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results as judged by the investigator
* Any condition that is unstable or could affect the safety of the patient and their compliance in the study as judged by the investigator
* Patients using high doses of non-steroidal anti-inflammatory drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Radiation Dermatitis Grade | 3 months (during radiation therapy and one month after)
  objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/European Organization for Research and Treatment of Cancer (RTOG/EORTC)
Radiation Dermatitis Assessment | 3 months (during radiation therapy and one month after)
  radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS)
Objective measurement of trans epidermal water loss of the skin | 3 months (during radiation therapy and one month after)
  Tewameter TM 300 will be used to objectively assess the skin barrier function by measuring the trans epidermal water loss of the skin
Objective measurement of the skin hydration | 3 months (during radiation therapy and one month after)
  Corneometer CM825 will be used to objectively assess the skin barrier function by measuring the skin hydration
Objective measurement of degree of erythema of the skin | 3 months (during radiation therapy and one month after)
  Mexameter MX18 will be used to objectively measure the degree of erythema of the skin
Analyze the skin cytokine content of the irradiated and non-irradiated breast | 3 months (during radiation therapy and one month after)
  Collect skin tape samples of the irradiated and non-irradiated breast in order to analyze these samples on cytokines by ELISA

SECONDARY OUTCOMES:
VAS-score | 3 months (during radiation therapy and one month after)
  Evaluation of pain using a visual analogue scale (VAS)
Skin dex 16 | 3 months (during radiation therapy and one month after)
  Health-related quality of life measure specific to skin diseases (Skindex-16)
Satisfaction with therapy | 3 months (during radiation therapy and one month after)
  Self-report on the efficacy of and the global satisfaction with the management of radiodermatitis
moist desquamation | 3 months (during radiation therapy and one month after)
  Onset time of moist desquamation

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis, Hasselt

IPD SHARING:
Plan to Share IPD: Undecided